CLINICAL TRIAL: NCT02540200
Title: A Pilot Study for Efficacy of BST-CarGel as an Adjunct to Microfracture for the Treatment of Chondral Lesions of the Hip: a Case Control Study
Brief Title: Efficacy of BST-CarGel in Treating Chondral Lesions of the Hip
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never started, no longer funded
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Ivan Wong, MD, MD, Nova Scotia Health Authority
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSHA-RS/2016-118
Record Dates: First submitted 2015-08-24; First posted 2015-09-03 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Disorder of Hip Region
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard treatment (Active Comparator): The patients undergo standard bone marrow stimulation technique (i.e. microfracture) for the treatment of their chondral lesions of the hip. This is currently the standard treatment for this condition.
  Interventions: Procedure: Microfracture
- BST-CarGel (Experimental): In addition to undergoing the standard intervention with microfracture, BST-CarGel (the device of interest for the study) is applied during the intervention.
  Interventions: Device: BST-CarGel; Procedure: Microfracture

INTERVENTIONS:
Device: BST-CarGel — BST-CarGel is a scaffolding material after microfracture treatment is performed in order to treat the chondral lesions. It assists in the repair process by stabilizing the clot in the cartilage lesion via adhesion and inhibition of clot retraction.
  Arms: BST-CarGel
Procedure: Microfracture — It is a bone marrow stimulation technique, and the standard treatment for chondral lesions of the hip joint.

SUMMARY:
Hip pain in young patients is difficult to diagnose and treat. However, with advanced imaging techniques and surgical method, the investigators are able to identify hip cartilage lesions as a cause for the hip pain. MR (magnetic resonance) arthrography is the best imaging modality to diagnose chondral lesions of the hip, but it occasionally miss the pathology, thus necessitating a more accurate and invasive means of diagnosis. Consequently, hip arthroscopy is increasingly used for both diagnosis and treatment for hip cartilage pathology.

Microfracture is a means of stimulating bone marrow, and is a standard treatment for small chondral lesions. This procedure has shown to result in excellent functional and anatomical outcomes. Microfracture is now recognized as a standard treatment for cartilage lesions in the knee, and recently the indications of this technique extended to hip pathology.

The BST-CarGel device (Piramal Life Sciences, Bio-Orthopaedic Division) is based on the patented technology for cartilage repair. BST-Gel comprised of the buffer beta-glycerophosphate and chitosan, which is a well-studied natural material that is biocompatible and appropriate for its use as a scaffold to assist in cartilage repair. BST-Gel is mixed with the patient's whole blood and delivered to a surgically prepared cartilage lesion in conjunction with bone marrow stimulation. The BST-CarGel/blood mixture solidifies in the cartilage lesion and provides a three-dimensional scaffold for the repair process. This product has shown to result in superior chondral lesion repair when compared to the bone marrow stimulation alone.

The current study will collect data through standard of care practice when BST-CarGel in conjunction with a bone marrow stimulation technique is used for the treatment of focal cartilage lesions in the hip. In addition, these patients in the study group will be compared with the group o patients who undergo the bone marrow stimulation technique alone. The efficacy of BST-CarGel in conjunction with microfracture for cartilage lesions in the knee has been shown in previous studies. Additional research is required to expand knowledge and develop treatment guidelines for the treatment of the cartilage lesions in the hip using BST-CarGel. As the BST-CarGel improves the results of the bone marrow stimulation techniques without increasing the risks of the procedure, this device can be very beneficial in the case of cartilage lesions in the hip.

DETAILED DESCRIPTION:
Osteoarthritis of the hip is a disabling condition which leads to tremendous burdens to the patients and the society. It is difficult to pinpoint the cause of osteoarthritis in most cases but it is thought to be multifactorial, with genetic, biomechanical, structural and morphological factors as main contributors. Early identification and intervention of the osteoarthritic hip had been challenging due to the lack of accurate diagnostic tools and effective methods of intervention. However, recent advancements of imaging modalities such as MR arthrography and increased use of arthroscopy have resulted in early identification of acetabular labral pathology which may contribute to the development of osteoarthritis. Femoroacetabular impingement (FAI) is a condition where abnormally shaped hip causes impingement symptoms with the functional range of the hip, leading to labral pathology. Consequently, FAI is a significant contributor to the development of hip osteoarthritis. However, diagnosis of FAI can often be challenging as some patients present with impingement symptoms without clear radiographic signs. Hip arthroscopy, therefore, remains the gold standard for diagnosing chondral lesions as it allows direct visualization. Consequently, young patients with hip pain without radiographic evidence would often undergo arthroscopy of the hip, which can not only identify the underlying pathology but also provide tools to treat the problems.

Microfracture is a standard treatment for small chondral defects with excellent results and low complication rates. This procedure leads to attraction of undifferentiated stem cells into the chondral defects. These cells are stabilized by a marrow clot and differentiate into stable fibrocartilaginous tissue. This technique has been studied much more extensively in the knee than in the hip, with excellent short-term and long-term results. Microfracture has shown to result in better functional outcomes compared to the autologous chondrocyte implantation, with an equivalent histological outcome. Success in this technique in the knee led to application of the same technique in the hip joint with excellent results. Philippon and the colleagues followed nine patients with full-thickness chondral defects who underwent microfracture via hip arthroscopy. Eight patients had 95% to 100% coverage of the chondral defects as seen in second look revision hip arthroscopy. In addition, the study by Karthikeyan and the colleagues showed that 19 out of 20 patients had the average fill of 96% when the chondral defects were treated with microfracture. Several studies have shown that this anatomic restoration translates into functional improvements as well. McDonald and the colleagues showed that professional hockey players who underwent microfracture for Outerbridge grade IV chondral lesions were able to return to competitive games without a statistically significant decrease in performance when compared to the matched control cohort. In addition, the study by Domb and the colleagues shows significant improvements in patient-reported outcomes at two year follow-ups for the patients who underwent arthroscopic hip surgery with a microfracture procedure. This successful transition has set the precedent for adapting the effective techniques and tools used in the knee to treat hip pathology.

However, the bone marrow stimulating technique alone was not the perfect solution for the focal chondral defects, and various techniques and devices have been utilized to improve the efficacy of the current bone marrow stimulating technique. Recently, gel-forming biopolymer has gained interests as a scaffolding material that can be injected into the site of microfracture to stabilize the clot and facilitate the cartilage repair. Chitosan is a natural polysaccharide composed of D-glucosamine and N-acetyl-D-glucosamine residues, which is biocompatible and biodegradable. It is also pH-dependent where it remains dissolved in solution up to a pH of 6.2, and forms a hydrated gel-like precipitate once pH exceeds 6.2. Chitosan also remains liquid in room temperature but solidifies to a gel-like state at body temperature, which makes it an excellent injectable material. It has been studied extensively as an effective scaffolding biomaterial with low toxicity and great adhesiveness to tissues.

BST-CarGel (Piramal Life Sciences, Bio-Orthopaedic Division) is an injectable chitosan-based medical device which is designed to be used in conjunction with the bone marrow stimulation technique. It is comprised of the buffer β-glycerophosphate and chitosan, which is in a liquid state in room temperature. It is missed with the patients' untreated whole blood, and delivered to a surgically prepared cartilage lesion where microfracture is already performed. The BST-CarGel and blood mixture then solidifies in the cartilage defect forming a three-dimensional scaffold for the repair process by stabilizing the clot in the cartilage lesion via adhesion and inhibition of clot retraction. The resulting gel implant facilitates the body's own healing response, potentially by enhancing the residency of wound healing factors found in the blood along with bone marrow-derived cells.

The safety and efficacy of BST-CarGel in treating chondral lesions in femoral condyles have been shown in a well-designed randomized, controlled trial by Stanish and the colleagues. In this study, BST-CarGel treatment in conjunction with the conventional bone marrow stimulation technique was superior to the microfracture alone in terms of lesion filling at 12 months period, with equivalent clinical benefits and safety profiles. The superiority in cartilage repair may imply improved long-term clinical outcomes although further studies are required to establish this correlation. BST-CarGel has received the European CE (Conformité Européenne) mark approval for the extended indication where it can be used in all synovial joints in Europe, although the clinical research on other joints is limited. BST-CarGel optimizes the result of bone marrow stimulation, as demonstrated by previous clinical results, without increasing the inherent risks for this type of procedures. Therefore, BST-CarGel could be very beneficial in the case of chondral lesions in the hip.

In addition, the purpose of the treatment of the chondral lesions is not only the anatomic restoration of the defect but mainly the improvement of the clinical symptoms. The conventional bone marrow stimulation technique via microfracture has shown to improve the patients' functional outcomes. The visual analogue scale (VAS) is a simple and valid tool that is widely used to evaluate the patients' pain. In addition, there are several questionnaires that are specifically designed for hip pain. Non-arthritic hip score (NAHS) has been proven to be a valid tool without floor or ceiling effect in measuring the disability from non-arthritic hip pathology. International hip outcome score (iHOT) is a valid tool in measuring the patient-reported quality of life score. The original questionnaires which include 33 items are shown to be valid and reliable.

ELIGIBILITY:
Inclusion Criteria:

1. A body mass index less than or equal to 30 kg/m2
2. An age from 18 to 40 years
3. Alpha angle of > 55 degree on plain AP (anterior-posterior) pelvis radiograph.
4. The study patient agrees to follow the recommended physiotherapy program, including exercises to complete at home
5. The study patient has understood and signed the informed consent form approved by the Research Ethics Board prior to any study protocol evaluations and is committed to complete the study as defined in this protocol and in the study patient's informed consent form.
6. MRI-identified delamination will be included in the CarGel group
7. Lesion size greater than 2cm2 on the intraoperative measurement.

Exclusion Criteria:

1. Any medical conditions which in the opinion of the investigator, makes the study patient unable to complete the study or is likely to interfere with the assessment of safety and efficacy of the BST-CarGel medical device
2. Any coagulation disorders of the blood or those receiving anticoagulant therapy
3. Rheumatoid arthritis, osteoarthritis and crystal arthropathies such as gout, pseudogout, etc., and any arthritic changes of the joint
4. Chondral damage opposing the cartilage lesion (kissing lesions)
5. Known allergy to chitosan or known hypersensitivity to crustaceans such as shrimp, lobster and crab
6. Any general pathology that might prevent the collection of data on an extended duration.
7. Grade 2 or higher chondral changes in intraoperative findings

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Safety (any potential side effects) | Patients will be followed up for a total of 1 year after the operation, and any potential side effects will be recorded and reviewed

SECONDARY OUTCOMES:
Lesion repair outcome (amount of repair measured on the MRI or magnetic resonance imaging) | MRI will be performed at 1 year post-intervention
VAS - Visual Analog Pain Score | Patients will fill out the questionnaires at 1 month, 6 months, and 12 months post-intervention during their clinic visit
NAHS - Non Arthritic Hip Score | Patients will fill out the questionnaires at 1 month, 6 months, and 12 months post-intervention during their clinic visit
iHOT-33 - International Hip Outcome Tool | Patients will fill out the questionnaires at 1 month, 6 months, and 12 months post-intervention during their clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Wong, MD, Principal Investigator — Nova Scotia Health Authority

IPD SHARING:
Plan to Share IPD: No